CLINICAL TRIAL: NCT03672643
Title: AN OPEN-LABEL, SINGLE-ARM STUDY OF THE LONG-TERM SAFETY OF XALKORI (REGISTERED) IN PATIENTS FROM CHINA WITH ADVANCED NON-SMALL CELL LUNG CANCER (NSCLC) HARBORING A TRANSLOCATION OR INVERSION EVENT INVOLVING THE ANAPLASTIC LYMPHOMA KINASE (ALK) OR ROS1 LOCUS WHO HAVE PREVIOUSLY BEEN TREATED ON A STUDY OF XALKORI (REGISTERED)
Brief Title: Long Term Safety Observation of Crizotinib in Chinese NSCLC Population
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial is terminated based on business decision, not due to safety concerns or regulatory requirements.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A8081067
Record Dates: First submitted 2018-07-19; First posted 2018-09-14 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-09

CONDITIONS: ALK or ROS1-positive NSCLC
Keywords: NSCLC
MeSH Terms: interventions — Crizotinib

STUDY DESIGN:
Intervention Model Description: single arm, open label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): Crizotinib
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — receive crizotinib orally
  Other Names: Xalkori

SUMMARY:
This study is to allow access to crizotinib who were treated in previous Pfizer-sponsored studies in China.

DETAILED DESCRIPTION:
This study is a phase 4 study, to continually access Xalkori to Chinese patients who were recruited in previous studies of Crizotinib in China, and only collect the safety data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were enrolled and treated in Studies A8081005, A8081007, A8081014, A8081029, or A8081063 and are still receiving crizotinib treatment at the time of enrollment into this study. OR Patients randomized to the chemotherapy arm in Studies A8081014 or A8081029 who have experienced investigator assessed disease progression and have not yet crossed over to receive crizotinib treatment.
2. No ongoing NCI CTCAE Grade 3 or intolerable Grade 2 adverse events considered to be related to crizotinib treatment
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-3
4. Adequate organ function as defined by the following criteria

Exclusion Criteria:

1. Use of any anticancer drug subsequent to crizotinib prior to study entry
2. Use of drugs or foods that are known potent Cytochrome P450 (CYP)3A4 inhibitors
3. Use of drugs that are known potent CYP3A4 inducers
4. Concurrent use of drugs that are CYP3A4 substrates with narrow therapeutic indices, associated with life threatening arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- China (14):
  - Fujian Province Oncology Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Liwan District,Guangzhou, Guangdong
  - Eastern Theater General Hospital ,QinHuai District Medical Area, Nanjing, Jiangsu
  - Jilin Province Cancer Hospital, Changchun, Jilin
  - Jilin Provincial Cancer Hospital, Changchun, Jilin
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Sichuan Province Cancer Hospital/Department of Pulmonary Tumor, Chengdu, Sichuan
  - Sichuan Province Cancer Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Department of Respiratory, The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Internal Department, Beijing
  - Zhongshan Hospital Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
Supporting Information: Study Protocol, SAP, ICF, CSR
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A8081067

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 41 Chinese participants who were previously recruited in Pfizer-sponsored Crizotinib studies (A8081005 [NCT00932451], A8081014 [NCT01154140], A8081029 [NCT01639001], A8081063 [NCT01945021]) were enrolled in the current study to continue treatment with Crizotinib.
Groups:
- Crizotinib: Participants received Crizotinib 250 milligrams (mg) orally twice daily (BID) administered in treatment cycle of 28 days until disease progression, unacceptable toxicity, consent withdrawal, or death, whichever occurred first.
Period: Overall Study
Arm/Group | Crizotinib
Started | 41
Completed | 0
Not Completed | 41
Not completed — Adverse Event | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Not completed — Progressive disease | 11
Not completed — Global deterioration of health status | 1
Not completed — Refused further treatment | 7
Not completed — Rolled over to a continuous study for Crizotinib treatment | 16

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who had been enrolled in the study, regardless of whether treatment was received.
Groups:
- Crizotinib: Participants received Crizotinib 250 mg orally BID administered in treatment cycle of 28 days until disease progression, unacceptable toxicity, consent withdrawal, or death, whichever occurred first.
Arm/Group | Crizotinib
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 41
  Ethnicity: Not Hispanic or Latino | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 or 4 Adverse Events (AEs), Grade 5 AEs, AEs Lead to Treatment Discontinuation, Serious AEs (SAEs)- All Causality: Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03
Description: An AE was any untoward medical occurrence in a clinical study participant associated with the use of study intervention, whether or not considered related to the study intervention. According to NCI CTCAE version 4.03: Grade 3 indicates severe AE, Grade 4 indicates life-threatening consequences and urgent intervention indicated and Grade 5 indicates death related to AE. Participants who discontinued treatment due to AEs were captured under AEs leading to treatment discontinuation. SAE was any untoward medical occurrence at any dose that resulted in death; life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect or that was considered as an important medical event.
Time Frame: From first dose of study treatment up to 28 days after last dose (maximum follow up approximately up to 52.3 months; maximum exposure to treatment was 51.3 months)
Population: Safety analysis set included all participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib
Number analyzed (Participants) | 41
Participants
  Grade 3 or 4 AEs | 19
  Grade 5 AEs | 2
  AEs Leading to Treatment Discontinuation | 4
  SAEs | 13

2. Primary Outcome: Number of Participants With Grade 3 or 4 AEs, Grade 5 AEs, AEs Leading to Treatment Discontinuation and SAEs- Treatment Related: Assessed by NCI CTCAE v4.03
Description: An AE was any untoward medical occurrence in a clinical study participant associated with use of study intervention, whether or not considered related to study intervention. AEs that were related to treatment were evaluated in this outcome measure. Treatment relatedness was judged by investigator. According to NCI CTCAE version 4.03: Grade 3= severe AE, Grade 4= life-threatening consequences and urgent intervention indicated, Grade 5= death related to AE. Participants who discontinued treatment due to treatment related AEs were captured under AEs leading to treatment discontinuation. SAE was any untoward medical occurrence at any dose that resulted in death; life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect or that was considered as an important medical event.
Time Frame: as for outcome 1
Population: Safety analysis set included all participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib
Number analyzed (Participants) | 41
Participants
  Treatment Related Grade 3 or 4 AEs | 11
  Treatment Related Grade 5 AEs | 0
  Treatment Related AEs Leading to Treatment Discontinuation | 1
  Treatment Related SAEs | 4

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 28 days after last dose (maximum follow up approximately up to 52.3 months; maximum exposure to treatment was 51.3 months)
Description: Same event may appear as both non-SAE and SAE, but what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Safety analysis set was evaluated.
Arm/Group | Crizotinib
All-Cause Mortality (participants affected / at risk) | 3/41
Serious Adverse Events (participants affected / at risk) | 13/41
Other Adverse Events (participants affected / at risk) | 8/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib (N=41)
Crohn's disease (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 2
Anal abscess (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Pyelonephritis chronic (Infections and infestations) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 1
Biochemical pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib (N=41)
Neutrophil count decreased (Investigations) | 8
White blood cell count decreased (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT03672643/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT03672643/SAP_001.pdf